CLINICAL TRIAL: NCT04462913
Title: Biometric Recognition and Rehabilitation Assessment of Lower Extremity Sports Injury Based on Gait Touch Information
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: OR001
Record Dates: First submitted 2020-06-29; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-06

CONDITIONS: Sport Injury; Osteoarthritis, Knee
Keywords: sports injury; gait touch information; machine learning
MeSH Terms: conditions — Osteoarthritis, Knee; Athletic Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Healthy control: According to the previous clinical diagnosis, volunteers who has never suffered the lower extremity sports injuries.
  Interventions: Other: no intervention
- Patients with sports injuries: According to the previous clinical diagnosis, patients who has suffered the sports injuries(including hip, knee, and ankle joint diseases).
  Interventions: Other: no intervention
- Patients with degenerative osteoarthritis: According to the previous clinical diagnosis, patients who has suffered the degenerative osteoarthritis.
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — This is an observation study, with no intervention

SUMMARY:
The current common clinical methods cannot truly reflect the biomechanical status of the knee joint. Based on the foot-knee coupling mechanism, the simple and practical dynamic gait touch information provided by the 3D force platform are closely related to the knee biomechanics. The purpose of this study is to investigate the disease feature recognition, computer-aided diagnosis and rehabilitation assessment based on the gait touch information related to lower limb injuries.

DETAILED DESCRIPTION:
Background:

The current common clinical methods cannot truly reflect the biomechanical status of the knee joint. The three-dimensional gait analysis is the gold standard, but it is difficult to apply clinically. There is an urgent need for a clinically practical method to quantitatively evaluate the biomechanics of the knee joint under dynamic weight bearing.

Methods:

50 healthy volunteers, 450 sports injuries patients (including hip, knee, and ankle joint diseases) and 50 patients with degenerative osteoarthritis were recruited.

55 passive reflective markers were placed bilaterally on the body. Lower extremity kinematics and dynamic plantar pressure during walking, jogging were collected.

Outcome evaluation indicators and statistical methods: The following indicators use repeated measurement two-factor analysis of variance: the left and right sides, different rehabilitation times are used as repeated measurement variables, to analyze the biomechanical changes of the lower limb joint biomechanics and gait touch information. A variety of machine learning methods (such as PCA, SVM, CNN, etc.) are used to analyze, and select the appropriate algorithm and parameters according to the learning effect. Finally, this study will establish a machine learning models for computer-aided diagnosis, treatment, and rehabilitation assessment.

ELIGIBILITY:
Inclusion Criteria:

* patients with a certain sports injury (soft tissue injury or degenerative osteoarthritis) of a joint of the lower limb (hip or knee or ankle or foot).

Exclusion Criteria:

* Cognitive impairment
* other injuries affecting movement performance.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Inclusion: one healthy control group: healthy volunteers; and patients with a certain sports injury (soft tissue injury or degenerative osteoarthritis) of a joint of the lower limb (hip or knee or ankle or foot).
  Exclusion: Cognitive impairment or other injuries affecting movement performance.
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2017-07-28 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
walking speed | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking.
ground reaction force | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking.
knee flexion angle | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking.
the moment of knee extension in the gait cycle | On the day of enrollment.
  Three-dimensional gait analysis system and plantar pressure were used during walking.

SECONDARY OUTCOMES:
The International Knee Documentation Committee (IKDC) score | On the day of enrollment.
  The International Knee Documentation Committee (IKDC) score was used to evaluate the knee health.The patients completed score by themselves. The lowest score is 0 and the highest score is 100.

CONTACTS AND LOCATIONS:
Overall Officials: Hongshi Huang, Doctor, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No